CLINICAL TRIAL: NCT03084991
Title: OPTical Coherence Tomography IMAging in Patients With Acute myocardiaL Infarction During Primary PCI (OPTIMAL)
Brief Title: OPTical Coherence Tomography IMAging in Patients With Acute myocardiaL Infarction (OPTIMAL)
Acronym: OPTIMAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Yu Bo, Director,Principal Investigator, Clinical Professor, Harbin Medical University
Other Study IDs: Harbin OCT-Registry
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; NSTEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT group: 1500 AMI patients with OCT imaging guidance during PCI
- CAG group: 3000 AMI patients without OCT imaging guidance during PPCI

SUMMARY:
The purpose of the study is to investigate the clinical outcomes, safety and cost-effectiveness of intravascular OCT imaging in patients with acute myocardial infarction undergoing percutaneous coronary intervention (PCI). About 4500 patients with acute myocardial infarction (estimated 1500 with OCT guidance and 3000 without OCT guidance during PCI）will be prospectively enrolled in 20 sites in China. The total duration of the study is expected to be 5 years, 2 years for enrolment and 3 years for follow up.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry study of patients with acute myocardial infarction (AMI) that require catheterization. The purpose of this registry is to investigate the clinical outcomes, safety and cost-effectiveness of intravascular OCT imaging in patients with AMI undergoing PCI.The duration of the study is expected to be 5 years, 2 years for enrolment and 3 years for total follow up.The clinical study will be conducted in 20 centers in China.Approximately 4500 subjects (1500 with OCT imaging and 3000 without OCT imaging) will be enrolled in this study.Subjects will be followed up at 1, 3, 6, 12months and every 6 months afterwards up to 5 years. All subjects need to be followed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with:a.Symptoms of myocardial ischemia lasting for ≥ 30 minutes.b.Definite ECG changes indicating STEMI: ST elevation of greater than 0.1 mV in two contiguous limb leads or 0.2 mV in two contiguous precordial leads, or presumed new left bundle branch block. c. NSTEMI
* Referred for primary PCI.
* Are able to provide written Informed Consent prior to any study related procedure.

Exclusion Criteria:

* Patient who is unable to comply with the follow-up schedule.
* Left main occlusion
* Unable to restore TIMI flow grade III before stenting
* Prior coronary artery bypass surgery (CABG)
* Cardiogenic shock
* Patient who has any medical conditions that in the opinion of the investigator will not be appropriate to participate in the study.
* Patient has a life expectancy of less than 6 month due to any condition.
* Age ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMI who undergo primary PCI.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular adverse events rate | 1 year
  In patients treated conservatively, the safety objectives are to evaluate the occurrence of any adverse events in 1 year (re-infarction, re-hospitalization, revascularization by PCI or CABG, cardiac death, stoke, and major bleeding)

SECONDARY OUTCOMES:
The rate of procedural strategy changes during the primary PCI | baseline
  The rate of procedural strategy changes (thrombus aspiration or not, stenting or not, postdilation or not.) during the primary PCI.
The incidence of procedural complications | baseline
  The incidence of procedural complications including coronary artery dissection, acute occlusion, thrombosis, re-infarction, emergent coronary artery bypass graft, bleeding, no/slow reflow, and death.
the indience of different plaque characteristic in the setting of STEMI | baseline
  The incidence of plaque erosion, plaque rupture, calcified nodules, and other uncommon causes in the setting of STEMI.
Major cardiovascular adverse events rate | 2 and 3 year
  The incidence of major adverse cardiovascular events (MACE) at 24 months and 36 months after index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (20):
- China (20):
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Univerisity People'Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong general hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Guangxi medical university, Nanning, Guangxi
  - The Second Affiliated Hospital of Hebei Meidical University, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first affiliated hospital of Zhengzhou medical university, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The third hospital of Jilin University, Changchun, Jilin
  - the second affiliated hospital of Dalian medical university, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xian, Shanxi
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Derived] Wang N, Xu YS, Feng X, Zeng M, Chen X, Yu B, Kou JJ. Stress hyperglycemia ratio and long-term prognosis in patients with acute myocardial infarction undergoing percutaneous coronary intervention: evidence for an J-shaped association. J Geriatr Cardiol. 2025 Dec 28;22(12):981-991. doi: 10.26599/1671-5411.2025.12.001. PMID 41477146
- [Derived] Wang J, Fang C, Zhang S, Li L, Lu J, Wang Y, Wang Y, Yu H, Wei G, Yin Y, Jiang S, Guo J, Lei F, Liu H, Xu M, Ren X, Ma L, Tu Y, Xing L, Hou J, Dai J, Yu B. Systemic and local factors associated with reduced thrombolysis in myocardial infarction flow in ST-segment elevation myocardial infarction patients with plaque erosion detected by intravascular optical coherence tomography. Int J Cardiovasc Imaging. 2021 Feb;37(2):399-409. doi: 10.1007/s10554-020-02021-1. Epub 2020 Sep 28. PMID 32989612